CLINICAL TRIAL: NCT04888533
Title: Predicting Suicide: E.H.S.S.A. - An Efficient, Holistic, Heuristic and Semi-structured Suicide Assessment Tool for Accurately Predicting, in a Specific Patient, the Risk of Suicide in the Reasonably Foreseeable Future. (EHSSA)
Brief Title: Efficient, Holistic, Heuristic and Semi-structured Suicide Assessment Tool (EHSSA) - Very Accurate Prediction of Risk.
Acronym: EHSSA
Status: Completed | Type: Observational
Sponsor: Care Plus NJ, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: EHSSA prospective study- PESP
Record Dates: First submitted 2021-05-10; First posted 2021-05-17 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Suicide Risk
Keywords: Suicide Risk Assessment Tool; Holistic; Heuristic; Semi-structured; Predictive Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Patients evaluated by PESP during the trial period.: EHSSA tool applied to every patient in cohort.
  Interventions: Other: EHSSA- An Efficient and Holistic/Heuristic Semi-structured Suicide Assessment Tool

INTERVENTIONS:
Other: EHSSA- An Efficient and Holistic/Heuristic Semi-structured Suicide Assessment Tool — EHSSA will be used to evaluate every patient for suicide risk.
  Other Names: EHSSA

SUMMARY:
Many studies have found that insights regarding suicide risk-factors for cohorts does not translate to practical value in the identification of such risk in specific individuals.

E.H.S.S.A. - a suicide assessment tool that was empirically designed by an emergency psychiatry department (P.E.S.P. of Bergen County) in its effort to accurately predict, in specific patients, the risk of suicide attempts in the reasonably foreseeable future. It is of a unique paradigm that combines critical elements of holism, heuristics and semi-structured design.

DETAILED DESCRIPTION:
Objective:

Many studies have found that insight regarding suicide risk-factors for cohorts does not translate to practical value in the identification of such risk in specific individuals.

This performance improvement study formally examined the effectiveness of "EHSSA" (efficient, holistic/heuristic semi-structured suicide-risk assessment) - an empirically derived tool designed by this emergency psychiatry department. It is a suicide assessment tool for predicting in a specific patient (as opposed to a cohort), the risk of serious suicide attempts in the reasonably foreseeable future.

Methods:

At P.E.S.P. (Psychiatric Emergency Screening Program) of Bergen County of New Jersey, a prospective performance improvement study was done on all patients (N = 1,505) that had presented with psychiatric crisis to the department over the course of a 6 month period, (of which approximately 50% had significant suicidal ideations). The only exclusionary criteria was active delirium.

Each patient was evaluated using "EHSSA" by departmentally trained mental health professionals. Patients were deemed to either require hospitalization or be safe to be discharged to the community (with appropriate outpatient referrals). Those that were discharged (N = 137) were followed up with phone calls approximately 15 days post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age/gender/economic class with or without dementia and/or substance use disorders
* All patients presenting to P.E.S.P.(Psychiatric Emergency Screening Program of Bergen County) in psychiatric distress/crisis.

Exclusion Criteria:

- Active Delirium.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of any age/gender/economic class with or without dementia or substance use disorders who presented to the psychiatric emergency program (P.E.S.P.- Psychiatric Emergency Screening Program of Bergen County) in psychiatric distress/crisis during a discreet 6 month period.
Sampling Method: Non-Probability Sample
Enrollment: 1505 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Rate or number of completed or attempted suicide. | 6 months
  Reported/ascertained cases among the cohort of completed or serious suicide attempts within 15 days of EHSSA evaluation and discharge to community or until the start of treatment with an outpatient mental health professional, whichever came sooner.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kim, M.D., Principal Investigator — Care Plus NJ, Inc.
Locations (1):
- Care Plus NJ, Inc.- PESP (Psychiatric Emergency Screening Program), Paramus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided